CLINICAL TRIAL: NCT06762626
Title: A Randomized Controlled Trial Comparing Frozen Embryo Transfer Guided by Endometrial Receptivity Analysis Vs Standard Timing in Patients with Recurrent Implantation Failure
Brief Title: Comparing FET Guided by ERA Vs Standard Timing in Patients with Recurrent Implantation Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other); Kwong Wah Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Liuzhou Maternity and Child Healthcare Hospital (Other); Third Affiliated Hospital of Zhengzhou University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Professor Ernest Hung-Yu Ng, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HERA China
Record Dates: First submitted 2024-12-20; First posted 2025-01-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Implantation Failure; Infertility
Keywords: Endometrial receptivity analysis; ERA; RIF; Recurrent implantation failure; frozen embryo transfer; FET
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERA group (Experimental): The timing of frozen embryo transfer will be arranged according to the endometrial receptivity analysis result
  Interventions: Other: Frozen embryo transfer according to endometrial receptivity analysis result
- Control group (No Intervention): Frozen embryo transfer will be arranged according to standard timing, i.e. after 5 days of consecutive progesterone use

INTERVENTIONS:
Other: Frozen embryo transfer according to endometrial receptivity analysis result — Frozen embryo transfer will be arranged according to endometrial receptivity analysis result, which will be shown in the form of P+X hours
  Arms: ERA group

SUMMARY:
The pregnancy rate of in vitro fertilisation (IVF) remains around 35% per transfer. Women who are not pregnant following several embryo transfers are regarded as having recurrent implantation failure (RIF), with one of the causes being the asynchronization of the embryo and endometrium. Endometrial receptivity analysis (ERA) may identify the window of implantation and guide the timing of embryo transfer to improve the pregnancy outcomes. However, there is no randomized controlled trial on the clinical effectiveness of ERA in women with RIF.

This is a multicenter double-blind randomized controlled trial. All participants will have an endometrial biopsy for ERA in a standard hormonal treatment cycle. They will then be randomly assigned in the central laboratory into the intervention or control group in a 1:1 ratio. At the transfer cycle, participants in the intervention group will have frozen embryo transfer timed according to the results of ERA while those in the control group will have the transfer according to the standard timing. The primary outcome is the ongoing pregnancy rate at 10-12 weeks at their first frozen embryo transfer.

DETAILED DESCRIPTION:
Trial design This is a multicenter randomized double-blind controlled trial evaluating the clinical effectiveness of ERA-guided frozen embryo transfer in improving the pregnancy rate of infertile women with RIF. All participants will first undergo a biopsy cycle to obtain an endometrial biopsy for ERA and will then be randomly assigned into the intervention or control group. At the transfer cycle, participants in the intervention group will have frozen embryo transfer timed according to the ERA result while those in the control group will have frozen embryo transfer according to standard timing.

Screening, recruitment and consent Women with RIF will be recruited from 10 hospitals across China. Recurrent implantation failure is defined as failure to achieve pregnancy after three embryo transfer of both fresh and frozen embryos.3 The inclusion and exclusion criteria is summarized in Table 1.

Table 1. Inclusion and exclusion criteria Inclusion criteria

1. Women with RIF
2. Women aged < 40 years
3. Body mass index of women between 18.5 (inclusive) and 30 (exclusive) kg/m²
4. Women with at least one high quality frozen blastocyst (BB grade or above) and planning to undergo a single blastocyst transfer
5. Women who will give written informed consent

Exclusion Criteria

1. Women with recurrent pregnancy loss (3 or more biochemical or spontaneous miscarriages)
2. Either partner with known chromosomal abnormalities including balanced translocations
3. Women undergoing preimplantation genetic testing
4. Women with endometrial thickness < 7 mm in the IVF cycle
5. Women with a confirmed diagnosis of stage III-IV endometriosis or adenomyosis affecting uterine cavity morphology
6. Women with a confirmed diagnosis of antiphospholipid syndrome
7. Pathologies affecting the uterine cavity, including polyps, submucosal fibroids, intramural fibroids > 4 cm, or hydrosalpinx

Eligible women will be counselled for the nature, purpose, procedures, expected duration, potential risks and benefits, and any possible discomforts of the trial during recruitment. Participation is voluntary. All participants will be required to sign a written informed consent and no study-related procedure will be performed without any consent.

Demographic data of all participants will be recorded, which includes their age, height, weight, body mass index, smoking and education level. Their medical history and physical examination will also be recorded, including the indication for IVF, details of previous embryo transfer, obstetrics history, previous medical, surgery or infection history. The results of laboratory tests will also be recorded if available, which include basic endocrine tests such as serum anti-mullerian hormones level and thyroid function tests.

Biopsy cycle All participants will go through a biopsy cycle in a hormonal treatment cycle to obtain an endometrial sample for ERA testing. Oral estradiol (Estrofem, Novo Nordisk A/S, Bagsværd Denmark) 2mg three times a day will be started on the first or second day of their menstrual cycle for 10-15 days, with a maximum of 22 days. Then transvaginal ultrasound will be performed to measure the endometrial thickness and blood will be taken for serum estradiol and progesterone levels. When the endometrial thickness is ≥ 7mm, serum estradiol level is > 150 pg/ml (or 500 pmol/ml) and serum progesterone level is < 1 ng/ml (or 3.18 nmol/L), oral dydrogesterone (Duphaston, Abbott, Illinois, U.S.) 10mg three times a day and vaginal progesterone gel (Crinone 8%, Merck KGaA, Darmstadt, Germany) 90mg daily will be started within 24 hours in addition to oral estradiol.

An endometrial biopsy will be performed in the out-patient clinic after using progesterone for 5 consecutive days (120 + 3 hours) as the starting of progesterone P + 0. The endometrial sample will be sent to the central laboratory (Hangzhou Yizhen Medical Laboratory, China) for ERA testing.

Sample collection and delivery An endometrial biopsy will be performed with a pipelle provided in the ERA kit under aseptic technique. The plunge will be withdrawn to create a negative pressure and a piece of endometrial tissue will be collected from the fundus to the internal cervical os. A tissue sample of around 50 to 70 mg will be collected.

The endometrial sample will be immediately transferred to a cryotube containing 1.5ml of RNA-later stabilizer liquid, which prevents the RNA from degradation during transport to the laboratory. Excessive blood or mucus within the sample will be removed to avoid RNA degradation. The collection tubes containing endometrial samples will be shaken to ensure thorough mixing of RNA solution with the endometrial samples. After labelling, the endometrial samples in the collection tube will be stored at 4℃ in the refrigerator for at least 4 hours and then transported at room temperature to the central laboratory for ERA.

Endometrial receptivity analysis RNA-Seq high-throughput sequencing technology will be used to detect the expression of nearly 250 genes related to endometrial receptivity. The endometrial implantation window of the analyzed samples will be obtained by bioinformatics analysis.

Transfer cycle Participants will be requested to have the frozen embryo transfer within 1-3 months of the biopsy cycle. The frozen embryo transfer is performed in a hormonal treatment cycle using the same endometrial preparation regimen as the biopsy cycle. The timing of embryo transfer will be based on their group allocation. For participants in the intervention group, the timing of frozen embryo transfer will be arranged according to the ERA result. For those in the control group, frozen embryo transfer will be arranged according to standard timing, i.e. after 5 days of consecutive progesterone use. The best quality blastocyst will be thawed and transferred first.

Details of the transfer cycle will be recorded, including endometrial thickness measurement, serum progesterone level, start date and time of progesterone, embryo transfer date and time, fertilization method and the Gardner grading of the embryo.

Follow-up After 14 days of frozen embryo transfer, participants will have blood tests for serum beta human chorionic gonadotropin (β-hCG), estradiol and progesterone level. The study ends if the participants are not pregnant.

If the participant is pregnant, follow-up will continue until one week postpartum. Ultrasound findings on the number of fetuses and fetal heart status will be recorded at 5 weeks and 10-12 weeks post-embryo transfer. Antenatal complications, delivery details and neonatal information will also be recorded. The study ends after one week postpartum or if pregnancy loss occurs during the follow-up period.

Randomization and blinding Randomization Randomization will be performed in the Hangzhou Yizhen Medical Laboratory, China after receipt of the endometrial samples and before proceeding to ERA. Women will be randomly assigned to either the interventional group or the control group in a 1:1 ratio. Randomization will be stratified according to the centers and the age of women (<35 vs ≥35 years) using a random number table.16 Each woman will be included and randomized only once in the study.

Blinding This is a double-blind study and neither the participants nor researchers will be aware of the group allocation. Researches in each participating centre will be notified by the laboratory of the recommended time of embryo transfer for each participant. The report will state the following: "it is recommended that this woman undergoes frozen blastocyst transfer at P+X hours."

Unblinding Unblinding will occur when the participant has blood tests for β-hCG, estradiol and progesterone levels 14 days after embryo transfer. Both participant and researchers will be informed of the group assignment. Participants in the control group who do not conceive can opt to replace the remaining frozen blastocysts in subsequent cycles based on the ERA results.

Study outcome Primary outcome The primary outcome is the ongoing pregnancy rate defined as pregnancy with fetal pulsation at 10-12 weeks.

Secondary outcome Secondary outcomes are the endometrial receptivity status, the biochemical pregnancy rate, clinical pregnancy rate, biochemical miscarriage rate, early miscarriage rate, ectopic pregnancy rate and live birth rate. Their definitions are listed in Table 2. Obstetrics outcomes include the incidence of gestational diabetes mellitus, preeclampsia, placenta previa, placental abruption and the mode of delivery. Neonatal outcomes include the gestational age, birth weight, Apgar scores, preterm rate, malformation rate and neonatal mortality rate.

Sample size The primary outcome measure is the ongoing pregnancy rate, which is expected to be 35% in the intervention group and 25% in the control group. With a two-sided test level α = 0.05 and power (1-β) = 80%, using PASS15 software and based on Fisher's exact test, the calculated sample size is 660 women (330 in the intervention group and 330 in the control group). Considering a 10% dropout rate, a total sample size of 734 participants is required (367 in the intervention group and 367 in the control group).

Data analysis Full analysis set, per protocol set and safety analysis sets will be analyzed. Full analysis set refers to those who have received at least one test and at least one evaluation on effectiveness. Per protocol set refers to all cases in the full analysis set who have completed the protocol-specified cycles and had no major protocol violations. Safety set refers to those who received at least one test after enrollment and had at least one safety evaluation.

Count data will be presented as frequencies and percentages, while measurement data will be presented with mean, standard deviation, median, maximum and minimum. The primary and secondary outcomes among different groups will be directly compared.

The ongoing pregnancy rates among three groups will also be compared: transfer with adjusted timing based on ERA-nonreceptive results, transfer with standard timing based on ERA-receptive results and transfer with standard timing in women with ERA-nonreceptive results.

ELIGIBILITY:
Inclusion Criteria:

1. Women with recurrent implantation failure
2. Women aged < 40 years
3. Body mass index of women between 18.5 (inclusive) and 30 (exclusive) kg/m²
4. Women with at least one high quality frozen blastocyst (BB grade or above) and planning to undergo a single blastocyst transfer
5. Women who will give written informed consent

Exclusion Criteria:

1. Women with recurrent pregnancy loss (3 or more biochemical or spontaneous miscarriages)
2. Either partner with known chromosomal abnormalities including balanced translocations
3. Women undergoing preimplantation genetic testing
4. Women with endometrial thickness < 7 mm in the IVF cycle
5. Women with a confirmed diagnosis of stage III-IV endometriosis or adenomyosis affecting uterine cavity morphology
6. Women with a confirmed diagnosis of antiphospholipid syndrome
7. Pathologies affecting the uterine cavity, including polyps, submucosal fibroids, intramural fibroids > 4 cm, or hydrosalpinx

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 734 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 8-10 weeks after embryo transfer
  Pregnancy with fetal pulsation at 10-12 weeks

SECONDARY OUTCOMES:
Endometrial receptivity status | 4 weeks after endometrial biopsy
  Number of participants showing out of phase endometrium
Biochemical pregnancy rate | 14 days after embryo transfer
  Number of patients with serum β-hCG ≥ 25 mIU/ml 14 days after embryo transfer / Number of patients who underwent embryo transfer * 100%
Clinical pregnancy rate | At 5th week of pregnancy
  Number of patients with an intrauterine gestational sac on transvaginal ultrasound at the 5th week of pregnancy / Number of patients who underwent embryo transfer * 100%
Biochemical miscarriage rate | At 5th week of pregnancy
  Number of patients with serum β-hCG ≥ 25 mIU/ml at the 5th week of pregnancy but without a gestational sac on transvaginal ultrasound / Number of biochemical pregnancies * 100%
Early miscarriage rate | up to 13 weeks of pregnancy
  Number of spontaneous miscarriages of one or more gestational sacs before 13th week of pregnancy / Number of clinical pregnancies * 100%
Ectopic pregnancy rate | Till the end of pregnancy
  Number of patients with an extrauterine pregnancy diagnosed by ultrasound, surgery, or histopathology / Number of biochemical pregnancies * 100%
Gestational diabetes mellitus | Until one week postpartum
  Number of pregnant participants with gestational diabetes mellitus
Preeclampsia | Until one week postpartum
  Number of pregnant participants with preeclampsia
Placenta previa | Until one week postpartum
  Number of pregnant participants with placenta previa
Placental abruption | Until one week postpartum
  Number of pregnant participants with placental abruption
Mode of delivery | Until one week postpartum
  Number of delivery as vaginal, instrumental or caesarean section
Live birth rate | Until one week postpartum
  Number of live births after 28 weeks / Number of patients who underwent embryo transfer * 100%
Gestational age | Until one week postpartum
  The gestational age at birth
Birth weight | Until one week postpartum
  Birth weight of the fetus
Apgar scores | Until one week postpartum
  Apgar scores at 1 and 5 minutes
Preterm rate | Until one week postpartum
  Number of birth before 37 completed weeks of gestation
Malformation rate | Until one week postpartum
  Number of fetus with congenital malformation
Neonatal mortality rate | Until 28 days after delivery
  Number of the baby who die within 28 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Study Director — The University of Hong Kong; Song Quan, MD, Study Chair — Southern Medical University
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request after publication of the main results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the main results
Access Criteria: Reasonable request for academic purposes